CLINICAL TRIAL: NCT05586009
Title: Comparative Study of Different Doses of Magnesium as a Protective Agent in Cisplatin Induced Nephrotoxicity in Patients With Head and Neck Cancer
Brief Title: Comparative Study of Different Doses of Magnesium as a Protective Agent in Nephrotoxicity in Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mohamed saad saad younis, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35629/8/22
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cisplatin Adverse Reaction
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Active Comparator): (n=25): receive cisplatin with hydration 1000mg magnesium (8 Meq) intravenous infusion ( IVI ).
  Interventions: Drug: cisplatin with hydration magnesium
- Group 2 (Active Comparator): (n=25): receive cisplatin with hydration 2000mg magnesium (16 Meq) ( IVI ).
  Interventions: Drug: cisplatin with hydration magnesium
- Group 3 (Active Comparator): (n=25): receive cisplatin with hydration 3000 mg magnesium (32 Meq) ( IVI ).
  Interventions: Drug: cisplatin with hydration magnesium

INTERVENTIONS:
Drug: cisplatin with hydration magnesium — Optimal doses of magnesium in prevention cisplatin induced nephrotoxicity

SUMMARY:
The goal of this [ type of study: intervential study is to compare between different doses of magnesium to prevent cisplatin induced nephrotoxicity.] In 75 participant population with head and neck cancer recieved cisplatin it aims to answer are: • • optimal doses of magnesium as 3 groups each group take 1gm of magnesium then second group take 2gm of magnesium and finally third group take 3gm of magnesium Researchers will compare [ 3 groups ] to see if [ magnesium has effects in prevention cisplatin nephrotoxicity].

DETAILED DESCRIPTION:
This study aims to:

* Investigate the potential role of magnesium in prevention of cisplatin induced nephrotoxicity in patient with head and neck cancer.
* Determine the optimal dose of magnesium (Mg).

Study Design :

* This is a randomized, controlled, parallel, prospective clinical study included 75 patients with head and neck cancer presented and treated at Clinical Oncology Department Tanta University Hospital, Tanta.
* This study will be approved by Research Ethics Committee of Tanta University.
* Randamization will be carried out based on days of hospital admission.

Treatment Protocol :

• All patients will be scheduled to receive the standard treatment of head and neck cancer. Concurent chemo radio therapy (CCRT) consisting of radiotherapy, cisplatin (40mg / m²) by intravenous infusion) . This regimen will be repeated weekly for 7 cycles .

Patients will be classified into three groups:

* Group 1 (n=25): receive cisplatin with hydration 500 mg magnesium (8 Meq) .
* Group 2 (n=25): receive cisplatin with hydration 1000 mg magnesium (16 Meq).
* Group 3 (n=25): receive cisplatin with hydration 2000 mg magnesium (32 Meq). Blood and urine sample will be drawn before and after treatment (7 cycles ).

For all patients the following will be performed:

1. Full history and physical examination.
2. Demographic data (patient weight, ideal body weight (IBW) and Body surface area (BSA) determination).
3. Renal function testing ( blood urea nitrogen (BUN), serum creatinine (SrCr), BUN/SrCr ratio, estimated glomerular filtration rate (eGFR), sodium (Na) level and magnesium (Mg) level ).
4. Nephrotoxicity will be defined according to common terminology criteria for adverse events version 5.00 (CTCAE) (U.S. Department Of Health And Human Services.,2017).
5. Measuring health-related quality of life.
6. Laboratory, radiologically, and endoscopic examination for oncological diagnosis.
7. Estimation level of Urinary neutrophil gelatinase associated lipocalin (NGAL), Urinary kidney injury molecule - 1( KIM - 1) and Serum soluble Fasl at baseline and within five days of the last cisplatin dose administration.
8. Liver function tests (AST and ALT) before and after treatment (7 cycle).

Provision of Privacy :

* Privacy of all data is guaranated and there will be a file with code number for every patient and include all investigations.
* All patients will give their written informed consents.
* Data of all patients will be private and confidential.
* Any unexpected risks appeared during the course of the research will be reported to patients and ethical committee on time.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with head and neck cancer recieved cisplatin ECOG <2 eGFR>59 ml/min/1.73 Adequate hematological parameters

Exclusion Criteria:

* pregnant and lactating women Using of nephrotoxic drugs as NSAIDs Patients with hypersensitivity to any drug used Diabetic patients Patients with cardiovascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
75 patients received magnesium with Treatment related Adverse Events as Assessed by CTCAE v5.0 At the end of cycle 7 of chemotherapy (each cycle is 7days) | At the end of cycle 7 of chemotherapy (each cycle is 7days)
  Optimal doses of magnesium

SECONDARY OUTCOMES:
75 patients received magnesium and access change of biomarkers levels From Baseline in nephrotoxicity at the end of cycle 7 of chemotherapy (each cycle is 7days) | At the end of cycle 7 of chemotherapy (each cycle is 7days)
  Kim-1, NGAL, FasL and MDA

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Saad younis, Tanta, Gharbia Governorate, Egypt